CLINICAL TRIAL: NCT01684332
Title: Study of the Effects of Three Strawberry Jams, Differing in Carbohydrate and Antioxidant Content, on Postprandial Response in Healthy Subjects
Brief Title: Postprandial Response to Different Jams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Alfredo Martinez, Professor of Nutrition and Food Science, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UNAV-078-2010
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Postprandial; Hyperglycemia, Postprandial; Feeding Behaviors; Antioxidant; Lipid Profile
Keywords: Antioxidant; glucose metabolism; jam; polyphenols; postprandial; strawberry
MeSH Terms: conditions — Hyperglycemia; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Sugar (HS) (Experimental): Study of the postprandial effects after consuming 60g of strawberry jam with high sugar content
  Interventions: Other: Strawberry Jam
- Low Sugar (LS) (Experimental): Study of the postprandial effects after consuming 60g of strawberry jam with low sugar content
  Interventions: Other: Strawberry Jam
- Low Sugar + Antioxidant (LSA) (Experimental): Study of the postprandial effects after consuming 60g of strawberry jam with low sugar content and an antioxidant extract from strawberry pulp
  Interventions: Other: Strawberry Jam

INTERVENTIONS:
Other: Strawberry Jam

SUMMARY:
The aim of this study is to investigate the effects of an acute intake of three different types of strawberry jam, differing in the carbohydrates and antioxidants content, on postprandial glucose metabolism, lipid profile, antioxidant status and satiety indices, in healthy adults.

DETAILED DESCRIPTION:
Study Design: Randomized, postprandial, crossover, double-blind intervention with three arms.

Subjects: Sixteen healthy adults

Product studied: At each arm, participants consume 60g of strawberry jam:

* High-sugar jam (traditional; HS),
* Low-sugar jam (without added-sugar; LS),
* Low-sugar jam including antioxidant extract from strawberry pulp (LSA).

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women
* Normal weight or overweight (BMI between 18.5 and 29.9 kg/m2)
* Age between 20 and 50 years old.

Exclusion Criteria:

* To suffer from any chronic disease related to metabolism,
* To follow concomitant medications,
* To follow slimming treatments or hormone replacement therapy,
* To have any inability to perform the follow-up,
* Smoking,
* Known food allergies,
* Pregnancy, lactation or menopause

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Plasma malondialdehyde (MDA) postprandial measure | up to 120 minutes
  Plasma MDA measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam

SECONDARY OUTCOMES:
Serum glucose postprandial concentration | Baseline, 30, 60, 90 and 120 minutes
  Serum Glucose measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Serum insulin postprandial concentration | baseline, 30, 60, 90 and 120 minutes
  Serum insulin measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
HOMA insulin resistance index | Baseline, 30, 60, 90 and 120 minutes
  HOMA-IR calculated at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Serum total cholesterol postprandial concentration | Baseline, 30, 60, 90 and 120 minutes
  Serum total cholesterol measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Serum HDL-cholesterol postprandial concentration | Baseline, 30, 60, 90 and 120 minutes
  Serum HDL-cholesterol measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Serum LDL-cholesterol postprandial concentration | Baseline, 30, 60, 90 and 120 minutes
  Serum LDL-cholesterol calculated at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Serum Uric Acid postprandial concentration | Baseline, 30, 60, 90 and 120 minutes
  Serum Uric Acid measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Plasma Glutathione Peroxidase postprandial activity | Baseline, 30, 60, 90 and 120 minutes
  Plasma Glutathione Peroxidase activity measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam
Postprandial Plasma Total Antioxidant Capacity | Baseline, 30, 60, 90 and 120 minutes
  Plasma Total Antioxidant capacity measured at baseline and each 30 minutes during 2 hours after consuming 60 g of the experimental jam

CONTACTS AND LOCATIONS:
Overall Officials: J. Alfredo Martínez, PhD, Principal Investigator — University of Navarra; M. Ángeles Zulet, PhD, Study Chair — University of Navarra; Marta Cuervo, PhD, Study Chair — University of Navarra; Santiago Navas-Carretero, PhD, Study Chair — University of Navarra; Idoia Ibero-Baraibar, MsC, Study Chair — University of Navarra
Locations (1):
- Department of Nutrition, Food Science and Physiology, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Ibero-Baraibar I, Cuervo M, Navas-Carretero S, Abete I, Zulet MA, Martinez JA. Different postprandial acute response in healthy subjects to three strawberry jams varying in carbohydrate and antioxidant content: a randomized, crossover trial. Eur J Nutr. 2014 Feb;53(1):201-10. doi: 10.1007/s00394-013-0517-7. Epub 2013 Apr 4. PMID 23553051
- See also: University of Navarra — http://www.unav.es